CLINICAL TRIAL: NCT04206384
Title: Efficacy of Low-Frequency, High-Intensity Ultrasound for Reduction in Subdermal Adipose Layers
Brief Title: Low-Frequency, High-Intensity Ultrasound for Waist Circumference Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CAO Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 005-00036-8
Record Dates: First submitted 2019-12-17; First posted 2019-12-20 (Actual); Results first posted 2021-08-20 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Abdominal Subcutaneous Fat
Keywords: Ultrasound; Low-Frequency
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Single Treatment Group
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment group (Experimental): Each patient shall receive a total of 3 treatments. Each treatment shall consist of applying the ultrasound device for 30 minutes to the skin surface, working the device methodically over the abdominal area. The device shall be set at the maximum emission level, have an intensity of approximately 1.0 watt/cm^2.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultimate Contour Body Sculpting Device

SUMMARY:
This study evaluates the effectiveness and safety of externally applied lower frequency ultrasound to the waist/abdominal region of adults to achieve a reduction of fat cells/tissues below the skin, evidenced by a reduction in patient waist circumference.

DETAILED DESCRIPTION:
This study is to evaluate principally the effectiveness, and secondarily the safety, of external application of lower frequency ultrasound to the waist/abdominal region of adults to achieve a reduction of adipose cells/tissues in the subcutaneous region. The application of higher frequency (200kHz to 3MHz) ultrasound for this purpose has previously been demonstrated and such devices have received clearance for treatment in the United States. The question remains whether application of ultrasound at a lower frequency (35kHz to 45kHz) can achieve comparable results without introducing any new or elevated risks to the patient. This study will apply 3 treatments of the ultrasound energy and evaluate the change in patient's waist circumference, which would be evidence of reducing sub-cutaneous adipose cells/tissues.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or above 18
* Body Mass Index ≥ 25.

Exclusion Criteria:

* Age equal to or below 17.
* Body Mass Index < 25.
* Open sores, wounds, or otherwise compromised skin in the treatment area
* History of keloid formation, hypertrophic scarring, or abnormal/delayed wound healing.
* Known or suspected pregnancy, or active nursing.
* General systemic conditions of arteriosclerosis, anemia, aortic aneurysm, or hypertension.
* Liver conditions such as hyperlipidemia, hepatitis, liver disease, or abnormal liver function.
* Diabetes or blood-glucose sensitivity
* Any prior invasive cosmetic surgery to the waist or abdominal area, such as liposuction.
* Hernias or diastasis recti within the treatment area.
* Concurrent, or within the last 6 months, participation in any clinical trial for another device or drug.
* Existing bacterial or viral infections (influenza, rhinovirus, hepatitis, pneumonia, tuberculosis, and the like)
* Presence of acne vulgaris, herpes zoster, psoriasis vulgaris, or similar skin conditions in the treatment area.
* Any type of cosmetic treatment to the target area within the last 6 months.
* Implanted active medical device anywhere in the subject, or metallic or polymeric implants in the vicinity of the treatment area.
* Currently undergoing, or recently underwent, chemotherapy or radiation treatment.
* Per the investigator's discretion, any physical or mental condition which may compromise the patient's safety or welfare.
* Failure to complete the study as outlined.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Just the Right Cruves, Midvale, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group
Started | 52
Completed | 42
Not Completed | 10
Not completed — Withdrawal by Subject | 8
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 5
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 52
Waist Circumference [Mean (Standard Deviation); unit: Inches] | 40.95 (5.32)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 29.36 (4.23)

OUTCOME MEASURES:

1. Primary Outcome: Waist Circumference Change
Description: Change in measurable circumference of the patient's abdominal area from Baseline to immediately after the 4-week follow-up assessment (approximately 6 weeks from Baseline).
Time Frame: The difference between the circumference measurement immediately prior to the first treatment (Baseline) to immediately after the 4-week follow-up assessment (approximately 6 weeks from Baseline).
Population: Participants who completed treatment process and follow-up visits as described.
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | Treatment Group
Number analyzed (Participants) | 42
Inches | -2.03 (0.77)

2. Secondary Outcome: Number of Participants With Pain
Description: Incidence of pain during each application of the device and/or immediately following each application of the device (up to 15 minutes after use of the device ceased).
Time Frame: Assessed during and immediately after (up to 15 minutes after use ceased) each application of the device, and at 1 week, 4 weeks, and 12 weeks post-treatment.
Population: Assessment of participant during or after any treatment application.
Measure: Number; unit: participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 52
participants | 3

ADVERSE EVENTS:
Time Frame: Collection and follow-up occurred over a space of up to 8 weeks.
Description: No difference in definition. Event collection consisted of enquiring of the participant any observations following application of the device. Participants were to keep a study diary and document any observations. Investigator reviewed study diaries and identified any comments that constitute an adverse event.
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 17/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=52)
Ringing in the ears (Ear and labyrinth disorders) | 7 (7) — During application of the device, some participants reported hearing a ringing or buzzing in their ears, although the device or applicator handpiece were not generating an externally audible noise.
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Participant developed a rash a day after a treatment.
Constipation (Gastrointestinal disorders) | 1 (1) — Participant developed constipation 2 days after a treatment session.
Inflammation / Heat Sensation (Skin and subcutaneous tissue disorders) | 5 (5) — Participant indicated feeling heat at the application site and/or presented with redness or inflammation of the treatment site.
Fatty Urine (Renal and urinary disorders) | 1 (1) — Participant described seeing fatty or cloudy urine
Vertigo (Ear and labyrinth disorders) | 1 (1) — Participant complained of vertigo when getting up from the treatment table following use of the device.
Headache (Nervous system disorders) | 1 (1) — Participant described having a mild headache, the evening after a treatment.

LIMITATIONS AND CAVEATS:
Due to the coronavirus (COVID-19) pandemic, the planned 12-week follow-up was conducted virtually. This prevented capture of the primary measurement at this timepoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT04206384/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/84/NCT04206384/ICF_001.pdf